CLINICAL TRIAL: NCT01238653
Title: Feasibility of a Minimally Invasive Image-Guided Surgery System for Hepatic Procedures
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment with limited population for study parameters.
Sponsor: Pathfinder Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PTI-LC-2009-02
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Liver Cancer
Keywords: liver; cancer; tumor; Pathfinder
MeSH Terms: conditions — Liver Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was designed to confirm that the surgeon is able to perform accurate liver surface registration including standard liver features used as landmarks during a scheduled laparoscopic liver procedure. The hypothesis is that there will be no clinically relevant difference between the error measurements obtained during the laparoscopic procedures in this study when compared with those obtained during previous open liver registration studies.

The surface of the liver will be manually swabbed with the study tracked laparoscopic probe with landmarks noted during data collection. After registration of the liver is obtained, the registration points obtained during this procedure will be evaluated by the surgeon by moving the tracked laparoscopic probe over the liver surface and evaluating the location of the tracked laparoscopic probe displayed on the guidance system three dimensional (3D) image. The surgeon will accept or reject the registration accuracy.

DETAILED DESCRIPTION:
The Pathfinder System used during this study is used for data collection purposes only and is not used during the surgical procedure as an image guided system.

Preoperative computed tomography (CT) scans, obtained as standard of care, will be used to generate the image guided liver system 3D liver surface images used during the study.

During the laparoscopic procedure, the Pathfinder device will be inserted through the standard laparoscopic ports (5mm or 10mm) being used for the staging procedure.

A total study population will include 20 subjects that complete the laparoscopic procedure scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic procedure
* Had a preoperative CT image that includes the liver

Exclusion Criteria:

* Severe cirrhosis of the liver
* Kidney failure or dialysis
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any subject scheduled for a laparoscopic procedure where liver surface visualization and surface swabbing is feasible with standard port placement.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The number of accurate liver surface registrations obtained in the laparoscopic environment compared to accurate liver surface registrations obtained in open procedures | 30 days
  Subjects are followed for the study 30days (+/- 14 days) and are considered to have completed the study following this 30 day follow-up visit.
  The performance of accurate physical-to-image registrations obtained during laparoscopic procedures will be compared with open liver registrations obtained from previous validation studies during open liver procedures.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Geller, M.D., Principal Investigator — UPMC, Montefiore Hospital Liver Cancer Center
Locations (1):
- UPMC, Montefiore Hospital Liver Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Pathfinder Company Link — http://www.liversurgery.com